CLINICAL TRIAL: NCT01109212
Title: The Effects of the Association Bindarit + Irbesartan Versus Irbesartan Alone on Albuminuria on Patients With Diabetic Nephropathy. Placebo-controlled Study
Brief Title: The Effects of Bindarit in Diabetic Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 004SC06084; 2006-006191-38 (EudraCT Number)
Record Dates: First submitted 2010-04-08; First posted 2010-04-23 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Diabetic Nephropathy
Keywords: Type 2-Diabetic Nephrophaty; bindarit; albuminuria; MCP-1
MeSH Terms: conditions — Diabetic Nephropathies; Albuminuria | interventions — bindarit

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bindarit (Experimental): Patients treated with bindarit 2x300 mg bid plus irbesartan 2x150 mg once a day for 12 weeks
  Interventions: Drug: Bindarit
- Placebo (Placebo Comparator): patients treated with placebo 2 tablets bid plus irbesartan 2x150 mg once a day for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bindarit — dosage form:tablet dosage:2x300 mg frequency:b.i.d duration:12 weeks
  Other Names: AF2838
  Arms: Bindarit
Drug: Placebo — dosage form: tablet dosage: n.a. frequency: 2xplacebo b.i.d duration:12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether bindarit is effective to reduce albuminuria, compared to placebo, in nephropathic patients treated with irbesartan, as a background therapy.

DETAILED DESCRIPTION:
This is a pilot phase II, double-blind, multicentre, randomized, placebo-controlled, parallel groups study in patients with DN undergoing irbesartan therapy.

According to screening urinary albumin excretion, at baseline and before randomization, all patients will be categorized into 2 strata:

Stratum 1: microalbuminuria (20 to 200 μg/min, in at least 2 of 3 consecutive overnight urine samples collected at the screening) Stratum 2: macroalbuminuria (>200 μg/min, in at least 2 of 3 consecutive overnight urine samples collected at the screening).

Within each stratum, patients will be randomly allocated on a 1:1 basis to the 2 treatment arms (after one month induction period):

* bindarit 600MG twice a day
* placebo All patients will be treated with irbesartan 300 mg/day as background therapy. After 12 months of treatment albuminuria will be evaluated as primary endopoint.

ELIGIBILITY:
INCLUSION CRITERIA

* male and female patients with no limitation of race, aged 30 to 70 years;
* Type 2 diabetes defined as: > 30 years of age at diagnosis; insulin not required within 6 months of initial diagnosis; no history of diabetic ketoacidosis; currently treated with diet, oral hypoglycemics or insulin [Brenner 2000];
* microalbuminuria defined as urinary albumin excretion, 20 to 200 µg/min in at least 2 of 3 overnight urine samples or macroalbuminuria defined as urinary albumin excretion, > 200 µg/min in at least 2 of 3 overnight urine samples, confirmed in the baseline collection; should baseline albuminuria data not to be available, the patient may be conditionally treated;
* glycosylated haemoglobin (Hb A1c) <12% at Screening [Brenner 2000];
* serum creatinine ≤ 3 mg/dL at Screening;
* normotensive patients or hypertensive patients on stable antihypertensive therapy over the last 3 months and without specific contraindications to angiotensin antagonist therapy;
* female patients of childbearing potential required to have a negative pregnancy test and use an approved birth control method;
* patients legally able to give written informed consent to the trial (signed and dated by the patient).

EXCLUSION CRITERIA

Patients cannot enter the trial under the following circumstances:

* patients hypersensitive or allergic to ARBs or bindarit or its components, or with a positive history for drug allergy;
* Type 1 diabetes [Brenner 2000];
* history of non diabetic renal disease, including renal artery stenosis [Brenner 2000];
* history of heart failure before enrolment [Brenner 2000];
* acute myocardial infarction, coronary artery bypass grafting within the past one month [Brenner 2000];
* cerebral vascular accident or coronary angioplasty within the past six months month [Brenner 2000];
* Transient Ischemic Attacks (TIA) in the past 12 months [Brenner 2000];
* primary aldosteronism or pheocromocytoma [Brenner 2000];
* severe uncontrolled hypertension (sitting diastolic blood pressure > 115 and/or sitting systolic blood pressure> 220 mm Hg) in the previous 6 months;
* chronic use of corticosteroids, non-steroidal anti-inflammatory drugs, immunosuppressive drugs, MAO inhibitors;
* patients under the influence of alcohol or narcotics;
* patients treated with experimental drugs in the previous 4 weeks.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-03; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Urinary Albumin Excretion (µg/min) levels in the overnight urine specimen. | 12 weeks
  Relative change (per cent change) in Urinary Albumin Excretion (UAE) from the baseline

SECONDARY OUTCOMES:
Urinary Monocyte Chemoattractant protein (MCP-1/CCL2)(pg/ml) levels in the overnight urine specimen. | 12 weeks
  Relative change (per cent change) in Urinary MCP-1 levels from the baseline.
Serum lipids | 12 weeks
  Relative change (per cent change) in total cholesterol, cholesterol HDL, triglycerides, apolipoprotein-A, apolipoprotein-B from the baseline.
Safety and tolerability of bindarit in association of irbesartan. | 12 weeks
  Changes in anthropometrics, laboratory parameters and vital signs from the baseline. Number of adverse events.
Albuminuria remission rates | 12 weeks
  Rate of remission from macro to microalbuminuria and from micro to normoalbuminuria.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, PhD, Principal Investigator — Mario Negri Institute for Pharmacological Research
Locations (6):
- Italy (5):
  - Azienda Ospedaliera OO.RR. Bergamo - Unità Operativa Diabetologia, Bergamo, Bergamo
  - The Mario Negri Institute for Pharmacological Research- Clinical Research Center for Rare Diseases, Ranica, Bergamo
  - Azienda Ospedaliera di Treviglio-Caravaggio - Unità Operativa Malattie Metaboliche e Diabetologia, Treviglio, Bergamo
  - IRCCS Fondazione Centro S. Raffaele del Monte Tabor- Unità Operativa Medicina Generale, Milan, Milano
  - Ist. Patologia Medica e metodologia Clinica - Università di Sassari, Sassari, Sassari
- University Medical Center Dpt Endocrinology Diabetes and Metabolic Diseases- Diabetology Unit, Ljubljana, Ljubljana, Slovenia

REFERENCES:
- See also: Sponsor's website — http://www.angelinipharma.com